CLINICAL TRIAL: NCT04557670
Title: The Association Between Periodontal Health Status, Body Mass Index and Quality of Diet in a Sample of Adult Egyptian Patients. A Hospital Based Cross-sectional Study
Brief Title: Relationship Between Periodontal Health Status, Body Mass Index and Quality of Diet in a Sample of Adult Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, abdullah salem mohammed al-shantub, pricipal investigator, Cairo University
Other Study IDs: PER1-1-1
Record Dates: First submitted 2020-09-04; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Conditions Influencing Health Status

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a cross-sectional study investigating the relationship between periodontal health condition, body mass index and quality of diet on adult Egyptian dental patients attending the oral diagnostic center at faculty of Dentistry, Cairo University.

The faculty of Dentistry, Cairo University is an open public facility, a tertiary healthcare and a referral center

DETAILED DESCRIPTION:
* Dental patients will be recruited in a consecutive manner from the outpatient Diagnostic center, Faculty of Dentistry, Cairo University.
* Medical history will be taken, thorough oral examination will be done, and a full questionnaire will be filled for each patient.
* Before filling the questionnaire, the aim of the study will be explained to the patient and the patient's acceptance to participate in the survey will be received.
* Non-respondent patients or patients refusing to participate will be reported with the cause of their refusal.
* The questionnaire will be filled through a face-to-face personal interview with the patient using simple, short, easily comprehended questions.
* Full questionnaire will be filled, then full mouth periodontal examination and charting will be done for each patient.
* The interview questions will be prepared in English, translated into Arabic and then reverse translated by a certified translator to ensure accuracy.
* All the interviews will be done by the same investigator.
* Convetional Clinical examination will be held on a dental unit using the light of the unit and a mirror.
* Periodontal health status will be evaluated by full mouth charting using UNC 15 periodontal probe, including assessment of Probing Depth (PD), Clinical Attachment Level (CAL), Bleeding on probing (BOP), plaque index (PI), body mass index (BMI) and health eating index (HEI).
* The questionnaire which was applied in study will include the following:

  1. Questions including section for demographic information of age, gender, marital status, income, weight, length.
  2. Dietary habits were self-reported through completion of a short form of a validated food frequency questionnaire (Ruiz-Cabello et al., 2017).

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose age is between 18-70 years old.
2. Provide informed consent.
3. Patient have at least 20 natural teeth.
4. Patient had no received periodontal treatment within previous 4 months.

Exclusion Criteria:

1. Individuals with chronic systemic diseases such as cancer, osteoporosis, endocrine and hematological Pathologies.
2. Patients having problem in opening their mouth or undergoing inter-maxillary fixation where oral examination will not be possible.
3. Pregnant women.
4. Patients diagnosed with psychiatric problems or intoxicated with alcohol or drugs.
5. Patients with orthodontic appliances.
6. Patient had autoimmune condition.
7. All patients require prophylaxis at least those attending the diagnostic center.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult Egyptian dental outpatients attending the oral diagnostic center at faculty of Dentistry, Cairo University.
Sampling Method: Probability Sample
Enrollment: 328 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Periodontal health in association with Body mass index | An average of 1 year through study completion
  (weight and height will be combined to report BMI in kg/m^2)
  - To estimate the level of overweight and obesity. commonly used the (BMI); was calculated as the body weight (kg) divided by the square of the height (m^2).

SECONDARY OUTCOMES:
Quality of diet | An average of 1 year through study completion
  - Dietary habits were self-reported through completion of a short form of a validated food frequency questionnaire. in which participants indicated the frequency of consumption (number of times per day, week, month, or year) of 34 foods divided by food groups: fruit, vegetables, dairy products, fish, cereals, pulses, eggs, meat, fats, sweets, beverages, and nuts.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine-CU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No